CLINICAL TRIAL: NCT07035782
Title: Effect of Sevoflurane on Sweat Threshold in Children of Different Ages
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2025-03-214
Record Dates: First submitted 2025-04-13; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Child, Only; Temperature Regulation; Disorder; Low Body Temperatures; Sevoflurane
Keywords: Pediatric Anesthesia; Low Body Temperatures; Sevoflurane
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Birth to 28 days (Experimental): Children will undergo standard induction of sevoflurane anesthesia as described above, with body temperature monitored and sweating assessed using quantitative and qualitative methods
  Interventions: Device: temperature monitoring; Drug: Sevoflurane
- one month to 1 year (Experimental): Children will undergo standard induction of sevoflurane anesthesia as described above, with body temperature monitored and sweating assessed using quantitative and qualitative methods
  Interventions: Device: temperature monitoring; Drug: Sevoflurane
- 1 to 3 years (Experimental): Children will undergo standard induction of sevoflurane anesthesia as described above, with body temperature monitored and sweating assessed using quantitative and qualitative methods
  Interventions: Device: temperature monitoring; Drug: Sevoflurane
- 3 to 6 years (Experimental): Children will undergo standard induction of sevoflurane anesthesia as described above, with body temperature monitored and sweating assessed using quantitative and qualitative methods
  Interventions: Device: temperature monitoring; Drug: Sevoflurane
- 6 to 12 years (Experimental): Children will undergo standard induction of sevoflurane anesthesia as described above, with body temperature monitored and sweating assessed using quantitative and qualitative methods
  Interventions: Device: temperature monitoring; Drug: Sevoflurane

INTERVENTIONS:
Device: temperature monitoring — Core temperature will be measured in the distal esophagus. The esophageal probe will be inserted after intubation to the depth from the upper incisors recommended by Bloch et al,1 specifically one-quarter of the patient's height plus 4.5 cm.
Drug: Sevoflurane — Anesthesia induction will be standardized for all participants., the children will undergo inhalational induction using 8% sevoflurane with a fresh gas flow of 5 L/min in 100% oxygen. Once children loses consciousness, the sevoflurane concentration will be reduced to 3%-5% and then maintained as close as possible to 1.2 MAC, age-adjusted

SUMMARY:
Hypothermia is a common complication in pediatric anesthesia. Hypothermia will prolong the recovery time of anesthesia, and may also lead to increased oxygen consumption, prolonged blood coagulation time, and affect the metabolism of anesthetic drugs and postoperative immune function. Sevoflurane is the most commonly used inhaled anesthetic in children. This study explored the effect of sevoflurane on the sweat threshold of pediatric patients and analyzed the characteristics of body temperature regulation in children of different ages under anesthesia, which will help to understand the mechanism of body temperature regulation in children under anesthesia, and also provide a scientific basis for clinical anesthesia temperature management.

DETAILED DESCRIPTION:
Standardized anesthesia induction was used for all participants. The first step was mask oxygen inhalation under 5 L/min pure oxygen, and 8% sevoflurane was inhaled for induction. Once the child lost consciousness, the concentration of sevoflurane was reduced to 3%-5% and maintained at 1.2 MAC as much as possible. Tracheal intubation was then assisted with cisatracurium 0.2 mg/kg. Mechanical ventilation was maintained during the operation, and the end-tidal carbon dioxide level was monitored and maintained at about 35 mmHg. Caudal anesthesia with 0.25% ropivacaine was used to provide surgical site analgesia. TOF was performed throughout the procedure to monitor the depth of neuromuscular block. Core temperature was measured in the distal esophagus. The esophageal probe was inserted after intubation to a depth of one quarter of the patient's height plus 4.5 cm. Changes in surface humidity were monitored using an OM-62 humidity sensor, which was placed above the nipple line in the upper chest and suspended in the ostomy bag. The ostomy bag will be custom-cut as needed to ensure optimal fit and precise airflow control. Infants and young children (<6 years) will use a 4-cm diameter opening, while older children (6 to 12 years) will use a 6-cm diameter opening. To ensure smooth airflow in the stoma bag, a low flow meter will be used to accurately adjust the airflow rate to 0.5L/min. Skin water loss (in g/m²/h) will be calculated from airflow rate, temperature, and relative humidity, and sweating on the child's forehead will be observed and recorded every 3 minutes. The skin surface was wrapped with a plastic film to limit evaporation. An air mattress was used to cover the body up to the nipple line. Two disposable covers were placed on each chest and leg and connected to an inflatable heating device, respectively. The inflatable heating device was set to 43 ° C until the esophageal temperature reached 38 ° C. Core temperature as well as temperature and humidity in the ostomy bag were collected every minute. The Hotline system was used to warm the intravenous infusion. Once the patient's core temperature reached 38 ° C or the procedure was over, active warming was stopped. Heart rate and pulse oxygen saturation were continuously monitored, and blood pressure was measured every 3 minutes. Simulated data from the heart rate monitor, sweat sensor, respiratory gas monitor, and pulse oximeter were recorded at 3-min intervals using the data acquisition system described above. The end-expiratory anesthetic concentration during the whole procedure was also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 0-12 years old;
2. American Society of Anesthesiologists physical status I or II;
3. Weight within the normal range and body-mass index (BMI) for age between the 25th and 85th percentiles;
4. scheduled elective lower-body surgery under general anesthesia, expected to last at least 1 hour.

Exclusion Criteria:

1. The guardian of the child refused to participate in the study;
2. Operations involving extensive incisions, such as massive debridement or other operations requiring removal of large amounts of tissue;
3. Contraindications to esophageal temperature probe insertion (e.g., esophageal varices, congenital anomalies);
4. Thyroid dysfunction or autonomic dysfunction;
5. Premature infants (≤1 year old).

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The threshold esophageal temperature | During the operation
  The threshold esophageal temperature at which forehead sweating is first observed (any sustained increase in cutaneous water loss).

SECONDARY OUTCOMES:
The gain of sweating | During the operation
  the slope of the core temperature versus quantitative sweating rate from onset of sweating until the maximum is reached
Maximum sweating rate | During the operation
  as indicated by no further increase in sweat rate despite further increase in core temperature

CONTACTS AND LOCATIONS:
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University Wenzhou, Wenzhou, Zhejiang, China